CLINICAL TRIAL: NCT04113408
Title: MEningioma Detection Using Non Contrast MRI TecHniquEs
Acronym: MENTHE
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to lack of inclusion.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2019_15
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FABIR sequence — The FABIR sequence with a duration of 8 minutes is added to the imaging protocol.

SUMMARY:
Meningioma, an extra-axial brain tumor developed at the expense of meninges, accounts for 35% of central nervous system tumors, and its incidence is estimated at 3% in large autopsy series.

The current gold standard for screening and monitoring cerebral meningiomas is MRI with injection of gadoline-contrast product. However, the use of some of these products is problematic, due to gadolinium deposits observed in patients who have had several injections during their lifetime, especially in patients followed for multiple sclerosis.

Recently, the French National Agency for the Safety of Medicines and Health Products (ANSM) issued recommendations concerning the screening of meningiomas in patients at risk, particularly in people treated with cyproterone acetate. It is a synthetic progestogen steroid with anti-androgenic properties. It is used to treat hyperandrogenic syndromes in women or in the palliative treatment of prostate cancer in men. Its long-term use seems to be associated with a significant over-risk of developing meningiomas, brain tumours affecting meninges. This increased risk is multiplied by 7 in women exposed to high doses of cyproterone acetate, and by 20 over a cumulative dose of 60 grams, or about 5 years of treatment at 50 mg/day or 10 years at 25 mg/day. The ANSM recommends that a cerebral MRI be performed at the beginning of treatment for all patients, as well as a control MRI renewed at 5 years and then every 2 years if the MRI at 5 years is normal. These recommendations will lead to a large number of MRIs involving an injection of contrast agent in this population, with potential immediate or delayed serious adverse effects.

New techniques, such as Arterial Spin Labelling (ASL), or black blood sequences optimized for contrast detection, have been developed. These could detect meningeal anomalies and more particularly meningiomas without contrast injection, or with a significantly lower dose of contrast agent.

These techniques have not been specifically studied for screening or monitoring meningeal lesions, but it seems relevant and important to be able to validate protocols that reduce gadolinium doses given the high number of screening and follow-up MRIs in the general population.

Patients presenting for brain MRI for meningioma screening or follow-up will have the usual MRI sequences for their management, and the FABIR sequences without injection, added for research. These new sequences will add approximately 8 minutes of additional examination time.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient performing MRI as part of a screening or follow-up of known meningioma
* Express consent to participate in the study

Exclusion Criteria:

* Contraindication for MRI (electrical device, metallic foreign body, claustrophobia)
* Known hypersensitivity to the contrast medium (Gadolinium)
* Known renal failure: glomerular filtration rate <30mL/min
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the radiology department of the A. de Rothschild Foundation for an MRI, as part of a screening or monitoring of meningioma
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic concordance in terms of detection of cerebral meningiomas between the usual MRI sequences (Gold Standard) and the FABIR sequences without Gadolinium injection, performed as part of a meningioma screening or follow-up. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, Paris, France